CLINICAL TRIAL: NCT02670655
Title: Efficacy of Iontophoresis-assisted Ablative Fractional Laser Photodynamic Therapy With Short Incubation Time for the Treatment of Actinic Keratosis: 12-month Follow-up Results of a Prospective, Randomised, Comparative Trial
Brief Title: Efficacy of Iontophoresis-assisted AFL-PDT in Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Associate professor, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DAUderma-06
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Actinic Keratosis
Keywords: Ablative fractional laser; Iontophoresis; Actinic keratosis; Photodynamic therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Lidocaine; Prilocaine; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (short-time iontophoresis group) (Experimental): Group A was treated with iontophoresis-assisted AFL-PDT with a short incubation time (2 h)
  Interventions: Drug: lidocaine/prilocaine (5%) application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: MAL application; Device: Iontophoresis application; Device: irradiation with red light-emitting diode lamp
- Group B (short-time conventional group) (Active Comparator): Group B was treated with conventional AFL-PDT with a short incubation time (2 h)
  Interventions: Drug: lidocaine/prilocaine (5%) application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: MAL application; Device: irradiation with red light-emitting diode lamp
- Group C (long-time conventional group) (Active Comparator): Group C was treated with conventional AFL-PDT with a standard incubation time (3 h)
  Interventions: Drug: lidocaine/prilocaine (5%) application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: MAL application; Device: irradiation with red light-emitting diode lamp

INTERVENTIONS:
Drug: lidocaine/prilocaine (5%) application — For AFL pre-treatment, lidocaine/prilocaine (5%) cream (EMLA; Astra Pharmaceuticals, LP, Westborough, MA, USA) was applied to the treatment area under occlusion for 30 min
Device: 2940-nm Er:YAG AFL pretreatment — After the anaesthetic cream was removed, AFL therapy was performed using a 2940-nm Er:YAG AFL (Joule; Sciton Inc., Palo Alto, CA, USA) at 300-550 µm ablation depth, level 1 coagulation, 22% treatment density and a single pulse
Drug: MAL application — Immediately after AFL treatment, an approximately 1-mm-thick layer of MAL (Metvix, PhotoCure ASA, Oslo, Norway) was applied to the lesion and on 5 mm of surrounding normal tissue.
Device: Iontophoresis application — In Group A, ionotophoresis was performed on MAL-applied sites. We used iontophoresis (vitaliont II®, ITC Inc, Korea) with a patch. The active electrode was the anode, and 0.50-mA/cm2 current was applied to each AK lesion for 10 min.
  Arms: Group A (short-time iontophoresis group)
Device: irradiation with red light-emitting diode lamp — After incubation for 2 (Group A and B) or 3 hours (Group C), the dressing and cream were removed, and the area was cleansed with saline. The area was irradiated with a red light-emitting diode lamp (Aktilite CL 128; PhotoCure ASA, Oslo, Norway) with peak emission at 632 nm, placed 5 cm away from the skin surface, and a total light dose of 37 J/cm-2. All patients wore protective goggles during illumination.

SUMMARY:
Iontophoresis is a transdermal drug-delivery technique that enhances the transport of ionic species across membranes and may have significant benefit for the treatment of actinic keratosis (AK) by ablative fractional laser-primed photodynamic therapy (AFL-PDT).

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) with methyl-aminolevulinate (MAL) is effective in the treatment of actinic keratosis (AK). Many strategies have been studied to improve the production of protoporphyrin IX (PpIX), to improve efficacy of PDT. Pre-treatment of the skin with fractional laser resurfacing is a novel alternative technique to improve the efficacy of PDT for AK. Our previous studies showed that ablative fractional laser-primed PDT (AFL-PDT) offered higher efficacy than conventional MAL-PDT in the treatment of many diseases, such as AK, actinic cheilitis, Bowen's disease and basal cell carcinoma.1-4 Iontophoresis can be another method to improve efficacy of PDT. Iontophoresis is a transdermal drug-delivery technique which uses a mild electric current to enhance the transport of ionic species across membranes. Iontophoresis has been widely used to enhance drug delivery. Mizutani K et al.5 reported 5 AK patients successfully treated with direct-current pulsed iontophoresis-assisted 5-aminolevulinic acid (ALA)-PDT. Boddé HE et al.6 studied iontophoretic transport of ALA quantitatively in vitro and demonstrated enhanced transport of ALA by iontophoresis.

Until now, appropriate incubation time for AFL-PDT has not been elucidated. In our previous study, we investigated the efficacy of AFL-PDT with a short incubation time.7 Although AFL-PDT with a short incubation time (2 h) showed enhanced efficacy than conventional MAL-PDT with the standard incubation time, standard AFL-PDT with 3-h incubation time showed significantly higher efficacy than AFL-PDT with a short incubation time.

The aim of our study was to evaluate efficacy of iontophoresis in AFL-PDT for AK treatment. Consequently, we compared efficacy, recurrence rate, cosmetic outcome and safety between iontophoresis-assisted AFL-PDT with 2-h incubation time and conventional AFL-PDT with 2-h and 3-h incubation times.

ELIGIBILITY:
Inclusion Criteria:

* Korean patients aged ≥ 18 years who had biopsy-confirmed AK lesions

Exclusion Criteria:

* lactating or pregnant women
* patients with porphyria or a known allergy to any of the constituents of the MAL cream and lidocaine
* patients with systemic disease, history of malignant melanoma, tendency of melasma development or keloid formation, any AK treatment of the area in the previous 4 weeks, or any conditions associated with a risk of poor protocol compliance; and patients on immunosuppressive treatment
* metal-containing device (cardiac pacemaker, orthopaedic implants, gynaecological devices)
* cardiac arrhythmia
* large skin erosion

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Differences of short-term complete response rates between three groups | Short-term complete response rates were evaluated at 3 months
  The lesions were classified as either complete response (complete disappearance of the lesion) or incomplete response (incomplete disappearance of the lesion)
Differences of long-term complete response rates between three groups | Long-term complete response rates were evaluated at 12 months
  The lesions were classified as either complete response (complete disappearance of the lesion) or incomplete response (incomplete disappearance of the lesion)
Differences of recurrence rates between three groups | Recurrence rates were evaluated at 12 months
  In addition, the recurrence rate was evaluated 12 months after treatment. For the histopathologic evaluation of treatment response, at the 12-month follow-up visit, a 3-mm punch biopsy of the treated AK lesion was performed in all cases of clinically incomplete response.

SECONDARY OUTCOMES:
Differences of cosmetic outcomes between three groups | The overall cosmetic outcome was assessed 12 months after treatment
  Cosmetic outcomes were graded as excellent (slight redness or pigmentation change), good (moderate redness or pigmentation change), fair (slight-to-moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration)

OTHER OUTCOMES:
Difference of adverse events (erythema, post-inflammatory hyperpigmentation, edema, itching, oozing, bleeding) rates between groups | Within 12 months after each treatment
  Adverse events reported by the patient were noted at each follow-up visit, including severity, duration and need for additional therapy. All events due to PDT were described as phototoxic reactions (i.e., erythema, post-inflammatory hyperpigmentation, oedema, itching, oozing, bleeding and so forth).

IPD SHARING:
Plan to Share IPD: No